CLINICAL TRIAL: NCT02422901
Title: A Long-term Observational Study to Describe the Use of PASCORBIN® 7.5 g in Patients With Vitamin C Deficiency
Brief Title: A Long-term Study to Describe the Use of PASCORBIN® 7.5 g in Patients With Vitamin C Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 183A12VC
Record Dates: First submitted 2015-03-24; First posted 2015-04-22 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Vitamin C Deficiency; Acute Disease; Chronic Disease
MeSH Terms: conditions — Ascorbic Acid Deficiency; Acute Disease; Chronic Disease | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vit C deficiency in acute diseases: Patients with vitamin C deficiency due to a acute underlying disease treated with Pascorbin® 7.5 g
  Interventions: Drug: vitamin C
- Vit C deficiency in chronic diseases: Patients with vitamin C deficiency due to a chronic underlying disease treated with Pascorbin® 7.5 g
  Interventions: Drug: vitamin C

INTERVENTIONS:
Drug: vitamin C — According to the character of an observational study no intervention other than the administration of Pascorbin® 7.5g (which is administered routinely in these cases) is provided.
  Other Names: Pascorbin® 7.5g

SUMMARY:
The aim of this long-term observational study is the documentation of the use of PASCORBIN® 7.5 g in patients with vitamin C deficiency. Regarding the vitamin C deficiency, the investigators focus on the acquisition of data of the underlying diseases and the reduction of symptoms, that are related to oxidative stress and vitamin-C-deficiency. Next to this, exact assessment of medical tolerance and details of treatment requirements are further aims. Here the investigators take into account acute and chronic underlying medical conditions. Further health economic data are collected.

DETAILED DESCRIPTION:
The observational study began on 01 November 2012 and is scheduled for a period of 10 years continued (until 01 November 2022). The duration of the observational study for each patient is not fixed corresponding to the character of a non-interventional study. According to the underlying disease, characterized either acute or chronic, there are 2 and 3 observations within the treatment period, respectively. Documentation comprises the course of the underlying diseases (by tracking of general and diseases-specific symptoms), drug compatibility (by ADR assessment), concomitant medication or other treatment, health economic data, details of treatment regimen and standard epidemiological data.

ELIGIBILITY:
Inclusion Criteria:

* patients with vitamin C deficiency
* patients >= 12 years old

Exclusion Criteria:

* an oxalate urolithiasis,
* iron storage disorders (thalassemia, hemochromatosis, sideroblastic anemia) or have received recently transfused packed red blood cells
* under 12 years of age or
* are pregnant or breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a vitamin C deficiency due to acute or chronic underlying diseases
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-11; Primary Completion 2022-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change in general and disease-specific symptoms | therapy duration, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  The main aim was to measure the success of the treatment with Pascorbin® 7.5 g by the documentation of the change in general and disease-specific symptoms.
  The symptoms are measured by a score:
  0 = not present, 1 = slightly, 2 = moderate and 3 = strong
  The change of the symptoms is measured in change groups:
  * number of patients with improved symptoms
  * number of patients with unchanged symptoms
  * number of patients with worsened symptoms

SECONDARY OUTCOMES:
global assessment of efficacy of treatment with PASCORBIN® 7.5 g | therapy duration, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  Global assessment of efficacy is measured by a score:
  * Very good efficacy (complete regression of symptoms)
  * Good efficacy (symptoms was much improved)
  * Moderate efficacy (symptoms was slightly improved)
  * No efficacy (symptoms remained unchanged)
  * No efficacy (symptoms worsened)
Global assessment of tolerability of treatment with PASCORBIN® 7.5 g | on last visit, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  Global assessment of tolerability is measured by a score:
  * Very good tolerability (no side effects)
  * Poor tolerability (side effects occurred)
number of adverse reactions due to PASCORBIN® 7.5 g | on last visit, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  number of adverse reactions due to PASCORBIN® 7.5 g
epidemiology of the underlying diseases | on visit 1 (begin of the study) week 1
  number of patients with different underlying diseases due to vitamin C deficiency
therapy duration | time period between first and last infusion an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  measured in weeks or months
dosage scheme | therapy duration, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  number of infusions within the therapy duration

CONTACTS AND LOCATIONS:
Overall Officials: Holger Michels, MD & M. Sci., Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- multiple medical German Practices of physicians and medical practitioners, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
All data are anonymous. Patient data list only will be sent to regulatory authorities.

REFERENCES:
- [Derived] Vollbracht C, Raithel M, Krick B, Kraft K, Hagel AF. Intravenous vitamin C in the treatment of allergies: an interim subgroup analysis of a long-term observational study. J Int Med Res. 2018 Sep;46(9):3640-3655. doi: 10.1177/0300060518777044. Epub 2018 Jun 27. PMID 29950123